CLINICAL TRIAL: NCT05533671
Title: Conservative Versus Surgical Management of First Time Patella Dislocations
Brief Title: Conservative Versus Operative - First Time Patella Dislocations
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAU0964
Record Dates: First submitted 2022-09-04; First posted 2022-09-09 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Patella Dislocation
MeSH Terms: conditions — Patellar Dislocation

STUDY DESIGN:
Intervention Model Description: This study will be a prospective randomized controlled trial investigating outcomes (recurrent dislocation rates and participant reported outcomes) in two groups of participants following a primary patella dislocation. Half of the participants will be randomized to operative intervention with a standard medial patellofemoral ligament (MPFL) reconstruction and the other half will be randomized to conservative management with a standardized rehabilitation protocol (non-operative group).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Operative Group (Experimental): This group will have surgical procedure called a medial patellofemoral reconstruction where the kneecap is anchored back into its correct position)
  Interventions: Procedure: medial patellofemoral reconstruction
- Non-operative group (Active Comparator): This group will have physical therapy for their knee dislocation by following a specific rehabilitation plan.
  Interventions: Procedure: Non-operative group

INTERVENTIONS:
Procedure: medial patellofemoral reconstruction — Surgery to correct dislocated (knocked out of place) knee cap. This surgery anchors the kneecap back into the correct position and supports the kneecap.
  Arms: Operative Group
Procedure: Non-operative group — Physical therapy by following a specific regimen.
  Arms: Non-operative group

SUMMARY:
There is no consensus regarding whether rehabilitation or surgical management is best for the management of a primary patellar dislocation. Consequently this prospective randomized controlled aims to compare the incidence of recurrent knee dislocations and patient reported outcomes of patients with primary patellar dislocations managed with surgery (medial patellofemoral ligament reconstruction) compared to non-operative management (a standardized rehabilitation protocol, control group).

DETAILED DESCRIPTION:
Long term sequalae of first-time patellar dislocations include recurrent knee instability, osteoarthritis, and a decreased quality of life, and yet there is no consensus on the best management for these patients. Despite an increasing trend toward investigating operative vs non-operative management of primary patellar dislocations, scarce level-1 evidence exists comparing the two treatment modalities. Indeed, the few meta-analyses suggesting improved outcomes of operative treatment for first time patellar dislocations mainly utilize retrospective cohort studies. A randomized-controlled trial of 39 patients with primary patellar dislocations with a mean age of 24 (21 operative vs 18 non-operative), found decreased rates of recurrent knee instability after a mean follow up of 44 months (0% in operative vs 35% in non-operative), and a higher Kujala knee score (88.9 in operative vs 70.8 in non-operative; p=0.001). A controlled but non-randomized prospective controlled trial among 69 patients with a mean age of 18, (30 operative vs 39 non-operative), found lower rates of recurrent knee instability after a mean follow up of 24 months (0% in operative vs 20.5% in non-operative and a higher Kujala knee score (86.3 in operative group vs 80.03 in non-operative; p <0.05).The scarce randomized, prospective data investigating the appropriate management in primary patellar dislocations underscores the importance of the current study in providing high-quality evidence to the debate of how to best manage primary patellar dislocations. This study aims to compare the incidence of recurrent knee dislocations and patient reported outcomes of patients with primary patellar dislocations managed with surgery (medial patellofemoral ligament reconstruction) compared to non-operative management (a standardized rehabilitation protocol, control group).

ELIGIBILITY:
Inclusion Criteria:

* age 12 and older
* patients seen by the Columbia University Shoulder Elbow and Sports Medicine Service
* patients who experience a first-time patella dislocation

Exclusion Criteria:

* coexistent ligament injury or osteochondral fracture necessitating acute surgical intervention
* previous knee surgery
* knee instability prior to injury
* inability or unwillingness to adhere to study participate
* lost to follow up

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-09 (Estimated); Primary Completion 2032-09 (Estimated); Study Completion 2032-09 (Estimated)

PRIMARY OUTCOMES:
Change in Kujala Questionnaire Score at 2 weeks | Baseline and 2 weeks
  The Kujala questionnaire assess symptoms and limitations that a patient may experience as a result of a knee injury. Scores range from 0-100 with a higher score indicating less limitation. Scores will be reported at each time point.
Change in Kujala Questionnaire Score at 6 weeks | Baseline and 6 weeks
  The Kujala questionnaire assess symptoms and limitations that a patient may experience as a result of a knee injury. Scores range from 0-100 with a higher score indicating less limitation. Scores will be reported at each time point.
Change in Kujala Questionnaire Score at 3 months | Baseline and 3 months
  The Kujala questionnaire assess symptoms and limitations that a patient may experience as a result of a knee injury. Scores range from 0-100 with a higher score indicating less limitation. Scores will be reported at each time point.
Change in Kujala Questionnaire Score at 6 months | Baseline and 6 months
  The Kujala questionnaire assess symptoms and limitations that a patient may experience as a result of a knee injury. Scores range from 0-100 with a higher score indicating less limitation. Scores will be reported at each time point.
Change in Kujala Questionnaire Score at 1 year | Baseline and 1 year
  The Kujala questionnaire assess symptoms and limitations that a patient may experience as a result of a knee injury. Scores range from 0-100 with a higher score indicating less limitation. Scores will be reported at each time point.
Change in Kujala Questionnaire Score at 2 years | Baseline and 2 years
  The Kujala questionnaire assess symptoms and limitations that a patient may experience as a result of a knee injury. Scores range from 0-100 with a higher score indicating less limitation. Scores will be reported at each time point.
Change in Kujala Questionnaire Score at 5 years | Baseline and 5 years
  The Kujala questionnaire assess symptoms and limitations that a patient may experience as a result of a knee injury. Scores range from 0-100 with a higher score indicating less limitation. Scores will be reported at each time point.
Change in Kujala Questionnaire Score at 10 years | Baseline and 10 years
  The Kujala questionnaire assess symptoms and limitations that a patient may experience as a result of a knee injury. Scores range from 0-100 with a higher score indicating less limitation. Scores will be reported at each time point.
Time to first re-dislocation | Up to 10 years
  Time to first re-dislocation following intervention, measured in weeks

SECONDARY OUTCOMES:
Change in the Patient-Reported Outcome Measurement Information System (PROMIS) Physical Function (PF) at 2 weeks | Baseline and 2 weeks
  A computerized survey that asks a series of questions pertaining to a patient's physical function through a grading scale of activities of daily living. The Patient-Reported Outcome Measurement Information System (PROMIS) Physical Function (PF) computer adaptive test (CAT) is reported as a T-score with a mean of 50 and a standard deviation of 10. A higher score is indicative of a greater level of physical function.
Change in the Patient-Reported Outcome Measurement Information System (PROMIS) Physical Function (PF) at 6 weeks | Baseline and 6 weeks
  A computerized survey that asks a series of questions pertaining to a patient's physical function through a grading scale of activities of daily living. The Patient-Reported Outcome Measurement Information System (PROMIS) Physical Function (PF) computer adaptive test (CAT) is reported as a T-score with a mean of 50 and a standard deviation of 10. A higher score is indicative of a greater level of physical function.
Change in the Patient-Reported Outcome Measurement Information System (PROMIS) Physical Function (PF) at 3 months | Baseline and 3 months
  A computerized survey that asks a series of questions pertaining to a patient's physical function through a grading scale of activities of daily living. The Patient-Reported Outcome Measurement Information System (PROMIS) Physical Function (PF) computer adaptive test (CAT) is reported as a T-score with a mean of 50 and a standard deviation of 10. A higher score is indicative of a greater level of physical function.
Change in the Patient-Reported Outcome Measurement Information System (PROMIS) Physical Function (PF) at 6 months | Baseline and 6 months
  A computerized survey that asks a series of questions pertaining to a patient's physical function through a grading scale of activities of daily living. The Patient-Reported Outcome Measurement Information System (PROMIS) Physical Function (PF) computer adaptive test (CAT) is reported as a T-score with a mean of 50 and a standard deviation of 10. A higher score is indicative of a greater level of physical function.
Change in the Patient-Reported Outcome Measurement Information System (PROMIS) Physical Function (PF) at 1 year | Baseline and 1 Year
  A computerized survey that asks a series of questions pertaining to a patient's physical function through a grading scale of activities of daily living. The Patient-Reported Outcome Measurement Information System (PROMIS) Physical Function (PF) computer adaptive test (CAT) is reported as a T-score with a mean of 50 and a standard deviation of 10. A higher score is indicative of a greater level of physical function.
Change in the Patient-Reported Outcome Measurement Information System (PROMIS) Physical Function (PF) at 2 years | Baseline and 2 Years
  A computerized survey that asks a series of questions pertaining to a patient's physical function through a grading scale of activities of daily living. The Patient-Reported Outcome Measurement Information System (PROMIS) Physical Function (PF) computer adaptive test (CAT) is reported as a T-score with a mean of 50 and a standard deviation of 10. A higher score is indicative of a greater level of physical function.
Change in the Patient-Reported Outcome Measurement Information System (PROMIS) Physical Function (PF) at 5 years | Baseline and 5 Years
  A computerized survey that asks a series of questions pertaining to a patient's physical function through a grading scale of activities of daily living. The Patient-Reported Outcome Measurement Information System (PROMIS) Physical Function (PF) computer adaptive test (CAT) is reported as a T-score with a mean of 50 and a standard deviation of 10. A higher score is indicative of a greater level of physical function.
Change in the Patient-Reported Outcome Measurement Information System (PROMIS) Physical Function (PF) at 10 years | Baseline and 10 Years
  A computerized survey that asks a series of questions pertaining to a patient's physical function through a grading scale of activities of daily living. The Patient-Reported Outcome Measurement Information System (PROMIS) Physical Function (PF) computer adaptive test (CAT) is reported as a T-score with a mean of 50 and a standard deviation of 10. A higher score is indicative of a greater level of physical function.
Change in the Patient-Reported Outcome Measurement Information System (PROMIS) depression computer adaptive test (CAT) at 2 weeks | Baseline and 2 weeks
  A computerized survey that asks a series of questions pertaining to distress a patient may experience as a result of their injury, which can be followed over time to determine the effectiveness of an intervention. The Patient-Reported Outcome Measurement Information System (PROMIS) depression computer adaptive test (CAT) is reported as a T-score with a mean of 50 and a standard deviation of 10. A higher score is indicative of a greater level of depression.
Change in the Patient-Reported Outcome Measurement Information System (PROMIS) depression computer adaptive test (CAT) at 6 weeks | Baseline and 6 weeks
  A computerized survey that asks a series of questions pertaining to distress a patient may experience as a result of their injury, which can be followed over time to determine the effectiveness of an intervention. The Patient-Reported Outcome Measurement Information System (PROMIS) depression computer adaptive test (CAT) is reported as a T-score with a mean of 50 and a standard deviation of 10. A higher score is indicative of a greater level of depression.
Change in the Patient-Reported Outcome Measurement Information System (PROMIS) depression computer adaptive test (CAT) at 3 Months | Baseline and 3 Months
  A computerized survey that asks a series of questions pertaining to distress a patient may experience as a result of their injury, which can be followed over time to determine the effectiveness of an intervention. The Patient-Reported Outcome Measurement Information System (PROMIS) depression computer adaptive test (CAT) is reported as a T-score with a mean of 50 and a standard deviation of 10. A higher score is indicative of a greater level of depression.
Change in the Patient-Reported Outcome Measurement Information System (PROMIS) depression computer adaptive test (CAT) at 6 Months | Baseline and 6 Months
  A computerized survey that asks a series of questions pertaining to distress a patient may experience as a result of their injury, which can be followed over time to determine the effectiveness of an intervention. The Patient-Reported Outcome Measurement Information System (PROMIS) depression computer adaptive test (CAT) is reported as a T-score with a mean of 50 and a standard deviation of 10. A higher score is indicative of a greater level of depression.
Change in the Patient-Reported Outcome Measurement Information System (PROMIS) depression computer adaptive test (CAT) at 1 Year | Baseline and 1 Year
  A computerized survey that asks a series of questions pertaining to distress a patient may experience as a result of their injury, which can be followed over time to determine the effectiveness of an intervention. The Patient-Reported Outcome Measurement Information System (PROMIS) depression computer adaptive test (CAT) is reported as a T-score with a mean of 50 and a standard deviation of 10. A higher score is indicative of a greater level of depression.
Change in the Patient-Reported Outcome Measurement Information System (PROMIS) depression computer adaptive test (CAT) at 2 Years | Baseline and 2 Years
  A computerized survey that asks a series of questions pertaining to distress a patient may experience as a result of their injury, which can be followed over time to determine the effectiveness of an intervention. The Patient-Reported Outcome Measurement Information System (PROMIS) depression computer adaptive test (CAT) is reported as a T-score with a mean of 50 and a standard deviation of 10. A higher score is indicative of a greater level of depression.
Change in the Patient-Reported Outcome Measurement Information System (PROMIS) depression computer adaptive test (CAT) at 5 Years | Baseline and 5 Years
  A computerized survey that asks a series of questions pertaining to distress a patient may experience as a result of their injury, which can be followed over time to determine the effectiveness of an intervention. The Patient-Reported Outcome Measurement Information System (PROMIS) depression computer adaptive test (CAT) is reported as a T-score with a mean of 50 and a standard deviation of 10. A higher score is indicative of a greater level of depression.
Change in the Patient-Reported Outcome Measurement Information System (PROMIS) depression computer adaptive test (CAT) at 10 Years | Baseline and 10 Years
  A computerized survey that asks a series of questions pertaining to distress a patient may experience as a result of their injury, which can be followed over time to determine the effectiveness of an intervention. The Patient-Reported Outcome Measurement Information System (PROMIS) depression computer adaptive test (CAT) is reported as a T-score with a mean of 50 and a standard deviation of 10. A higher score is indicative of a greater level of depression.
Change in the Patient-Reported Outcome Measurement Information System (PROMIS) pain interference (PI) computer adaptive test (CAT) at 2 weeks | Baseline and 2 weeks
  A computerized survey that asks a series of questions pertaining to pain a patient may experience from an injury and the way it influences different domains of their life, which can be followed over time to determine the effectiveness of an intervention. The Patient-Reported Outcome Measurement Information System (PROMIS) pain interference (PI) computer adaptive test (CAT) is reported as a T-score with a mean of 50 and a standard deviation of 10.
Change in the Patient-Reported Outcome Measurement Information System (PROMIS) pain interference (PI) computer adaptive test (CAT) at 6 weeks | Baseline and 6 weeks
  A computerized survey that asks a series of questions pertaining to pain a patient may experience from an injury and the way it influences different domains of their life, which can be followed over time to determine the effectiveness of an intervention. The Patient-Reported Outcome Measurement Information System (PROMIS) pain interference (PI) computer adaptive test (CAT) is reported as a T-score with a mean of 50 and a standard deviation of 10.
Change in the Patient-Reported Outcome Measurement Information System (PROMIS) pain interference (PI) computer adaptive test (CAT) at 3 months | Baseline and 3 months
  A computerized survey that asks a series of questions pertaining to pain a patient may experience from an injury and the way it influences different domains of their life, which can be followed over time to determine the effectiveness of an intervention. The Patient-Reported Outcome Measurement Information System (PROMIS) pain interference (PI) computer adaptive test (CAT) is reported as a T-score with a mean of 50 and a standard deviation of 10.
Change in the Patient-Reported Outcome Measurement Information System (PROMIS) pain interference (PI) computer adaptive test (CAT) at 6 months | Baseline and 6 months
  A computerized survey that asks a series of questions pertaining to pain a patient may experience from an injury and the way it influences different domains of their life, which can be followed over time to determine the effectiveness of an intervention. The Patient-Reported Outcome Measurement Information System (PROMIS) pain interference (PI) computer adaptive test (CAT) is reported as a T-score with a mean of 50 and a standard deviation of 10.
Change in the Patient-Reported Outcome Measurement Information System (PROMIS) pain interference (PI) computer adaptive test (CAT) at 1 year | Baseline and 1 year
  A computerized survey that asks a series of questions pertaining to pain a patient may experience from an injury and the way it influences different domains of their life, which can be followed over time to determine the effectiveness of an intervention. The Patient-Reported Outcome Measurement Information System (PROMIS) pain interference (PI) computer adaptive test (CAT) is reported as a T-score with a mean of 50 and a standard deviation of 10.
Change in the Patient-Reported Outcome Measurement Information System (PROMIS) pain interference (PI) computer adaptive test (CAT) at 2 years | Baseline and 2 years
  A computerized survey that asks a series of questions pertaining to pain a patient may experience from an injury and the way it influences different domains of their life, which can be followed over time to determine the effectiveness of an intervention. The Patient-Reported Outcome Measurement Information System (PROMIS) pain interference (PI) computer adaptive test (CAT) is reported as a T-score with a mean of 50 and a standard deviation of 10.
Change in the Patient-Reported Outcome Measurement Information System (PROMIS) pain interference (PI) computer adaptive test (CAT) at 5 years | Baseline and 5 years
  A computerized survey that asks a series of questions pertaining to pain a patient may experience from an injury and the way it influences different domains of their life, which can be followed over time to determine the effectiveness of an intervention. The Patient-Reported Outcome Measurement Information System (PROMIS) pain interference (PI) computer adaptive test (CAT) is reported as a T-score with a mean of 50 and a standard deviation of 10.
Change in the Patient-Reported Outcome Measurement Information System (PROMIS) pain interference (PI) computer adaptive test (CAT) at 10 years | Baseline and 10 years
  A computerized survey that asks a series of questions pertaining to pain a patient may experience from an injury and the way it influences different domains of their life, which can be followed over time to determine the effectiveness of an intervention. The Patient-Reported Outcome Measurement Information System (PROMIS) pain interference (PI) computer adaptive test (CAT) is reported as a T-score with a mean of 50 and a standard deviation of 10.
Percentage of participants who re-dislocate their knee after treatment at each time point within each group | 2 weeks 6 weeks, 3 months, 6 months, 1 year, 2 years, 5 years and 10 years
  Percentage of group that experienced re-dislocation after treatment starts at each time point
Time to return to full activity or sports for each group | Up to 10 years
  Time from treatment initiation to full return to pre-injury activity levels in each group, measured in weeks
Change in the Banff Patella Instability Instrument at 2 weeks | Baseline and 2 weeks
  Quality of life survey developed in patients with patellofemoral instability that asks patients questions regarding how their patellofemoral injury has affected their life. it is on a scale of 0-100 with higher scores indicating better outcomes.
Change in the Banff Patella Instability Instrument at 6 weeks | Baseline and 6 weeks
  Quality of life survey developed in patients with patellofemoral instability that asks patients questions regarding how their patellofemoral injury has affected their life. it is on a scale of 0-100 with higher scores indicating better outcomes.
Change in the Banff Patella Instability Instrument at 3 months | Baseline and 3 months
  Quality of life survey developed in patients with patellofemoral instability that asks patients questions regarding how their patellofemoral injury has affected their life. it is on a scale of 0-100 with higher scores indicating better outcomes.
Change in the Banff Patella Instability Instrument at 6 months | Baseline and 6 months
  Quality of life survey developed in patients with patellofemoral instability that asks patients questions regarding how their patellofemoral injury has affected their life. it is on a scale of 0-100 with higher scores indicating better outcomes.
Change in the Banff Patella Instability Instrument at 1 year | Baseline and 1 year
  Quality of life survey developed in patients with patellofemoral instability that asks patients questions regarding how their patellofemoral injury has affected their life. it is on a scale of 0-100 with higher scores indicating better outcomes.
Change in the Banff Patella Instability Instrument at 2 years | Baseline and 2 years
  Quality of life survey developed in patients with patellofemoral instability that asks patients questions regarding how their patellofemoral injury has affected their life. it is on a scale of 0-100 with higher scores indicating better outcomes.
Change in the Banff Patella Instability Instrument at 5 years | Baseline and 5 years
  Quality of life survey developed in patients with patellofemoral instability that asks patients questions regarding how their patellofemoral injury has affected their life. it is on a scale of 0-100 with higher scores indicating better outcomes.
Change in the Banff Patella Instability Instrument at 10 years | Baseline and 10 years
  Quality of life survey developed in patients with patellofemoral instability that asks patients questions regarding how their patellofemoral injury has affected their life. it is on a scale of 0-100 with higher scores indicating better outcomes.
Change in Norwich Patellar Instability Score at 2 weeks | Baseline and 2 weeks
  Symptom survey that asks patients questions pertaining to symptoms they may be experiencing as a result of their knee injury. Scored as a percentage, a higher percentage indicates worse symptoms and therefore a worse outcome.
Change in Norwich Patellar Instability Score at 6 weeks | Baseline and 6 weeks
  Symptom survey that asks patients questions pertaining to symptoms they may be experiencing as a result of their knee injury. Scored as a percentage, a higher percentage indicates worse symptoms and therefore a worse outcome.
Change in Norwich Patellar Instability Score at 3 months | Baseline and 3 months
  Symptom survey that asks patients questions pertaining to symptoms they may be experiencing as a result of their knee injury. Scored as a percentage, a higher percentage indicates worse symptoms and therefore a worse outcome.
Change in Norwich Patellar Instability Score at 6 months | Baseline and 6 months
  Symptom survey that asks patients questions pertaining to symptoms they may be experiencing as a result of their knee injury. Scored as a percentage, a higher percentage indicates worse symptoms and therefore a worse outcome.
Change in Norwich Patellar Instability Score at 1 year | Baseline and 1 year
  Symptom survey that asks patients questions pertaining to symptoms they may be experiencing as a result of their knee injury. Scored as a percentage, a higher percentage indicates worse symptoms and therefore a worse outcome.
Change in Norwich Patellar Instability Score at 2 years | Baseline and 2 years
  Symptom survey that asks patients questions pertaining to symptoms they may be experiencing as a result of their knee injury. Scored as a percentage, a higher percentage indicates worse symptoms and therefore a worse outcome.
Change in Norwich Patellar Instability Score at 5 years | Baseline and 5 years
  Symptom survey that asks patients questions pertaining to symptoms they may be experiencing as a result of their knee injury. Scored as a percentage, a higher percentage indicates worse symptoms and therefore a worse outcome.
Change in Norwich Patellar Instability Score at 10 years | Baseline and 10 years
  Symptom survey that asks patients questions pertaining to symptoms they may be experiencing as a result of their knee injury. Scored as a percentage, a higher percentage indicates worse symptoms and therefore a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: David Trofa, MD, Principal Investigator — Associate Professor of Orthopaedic Surgery
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zheng X, Hu Y, Xie P, Cui M, Ma X, Feng YE, Gu J, Gao S. Surgical medial patellofemoral ligament reconstruction versus non-surgical treatment of acute primary patellar dislocation: a prospective controlled trial. Int Orthop. 2019 Jun;43(6):1495-1501. doi: 10.1007/s00264-018-4243-x. Epub 2018 Nov 20. PMID 30460463
- [Background] Xing X, Shi H, Feng S. Does surgical treatment produce better outcomes than conservative treatment for acute primary patellar dislocations? A meta-analysis of 10 randomized controlled trials. J Orthop Surg Res. 2020 Mar 24;15(1):118. doi: 10.1186/s13018-020-01634-5. PMID 32209111
- [Background] Liu Z, Yi Q, He L, Yao C, Zhang L, Lu F, Zhang X, Wu M, Geng B, Xia Y, Jiang J. Comparing Nonoperative Treatment, MPFL Repair, and MPFL Reconstruction for Patients With Patellar Dislocation: A Systematic Review and Network Meta-analysis. Orthop J Sports Med. 2021 Sep 28;9(9):23259671211026624. doi: 10.1177/23259671211026624. eCollection 2021 Sep. PMID 34604425
- [Background] Mackay ND, Smith NA, Parsons N, Spalding T, Thompson P, Sprowson AP. Medial Patellofemoral Ligament Reconstruction for Patellar Dislocation: A Systematic Review. Orthop J Sports Med. 2014 Aug 8;2(8):2325967114544021. doi: 10.1177/2325967114544021. eCollection 2014 Aug. PMID 26535352
- [Background] Bitar AC, Demange MK, D'Elia CO, Camanho GL. Traumatic patellar dislocation: nonoperative treatment compared with MPFL reconstruction using patellar tendon. Am J Sports Med. 2012 Jan;40(1):114-22. doi: 10.1177/0363546511423742. Epub 2011 Oct 19. PMID 22016458